CLINICAL TRIAL: NCT04177784
Title: Web Based Intervention to Reduce Weight Bias Among Dietitians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Emily Dhurandhar, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB2019-321
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Intervention Video (I); Weight Control Video (C1); Weight Neutral Control Video (C2)

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were told they would be participating in a study that aims to determine the effectiveness of online education in dietitians. They were unaware that determining the effect of the videos on weight bias was the objective of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (I) (Experimental): This arm was randomized to a 20 min video that emphasized information about factors other than individual behaviors that influence weight, weight loss and ability to maintain weight. It also indirectly addressed weight bias by explaining how to have conversation about weight and health with a patient with obesity that is free of biases.
  Interventions: Other: Online Educational Videos
- Weight Control (C1) (Active Comparator): This arm was randomized to a 20 min video that emphasized the controllable aspects of weight and gave dietitians an overview of a tool to help plan and monitor weight loss.
  Interventions: Other: Online Educational Videos
- Weight Neutral Control (C2) (Placebo Comparator): The arm was randomized to a 20 min video about the role dietitians play in society, that made no mention of weight or obesity.
  Interventions: Other: Online Educational Videos

INTERVENTIONS:
Other: Online Educational Videos — The videos were developed by the researchers based on a prior study to test if specific information about obesity and weight control influence weight bias.

SUMMARY:
Weight bias in dietitians is prevalent and may affect patient care. The investigators conducted a randomized controlled trial to test if explicit and implicit bias could be influenced by a short, 20 minute educational video.

DETAILED DESCRIPTION:
This randomized controlled trial studied the effect of three different videos on weight bias in a nationally representative sample of dietitians. The "intervention" group (I) watched a video about the etiology of obesity, reasons for weight regain, and how to talk to patients about weight. The first "control" group (C1) received information about the role of the environment and individual behavior in weight gain, and tools to help patients control their weight. The second control group (C2) received a weight neutral video about the role of dieticians in society. Bias measures were taken before and just after watching the video, and again one month later.

ELIGIBILITY:
Inclusion Criteria:

* Any dietitian in the Clinical Dietitian Registry Database.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Change in "Blame" explicit bias | Change from pre to immediately post intervention (1 hour)
  "Blame" subscore of Anti-fat Attitudes Test, higher score means more bias
Change in "Blame" explicit bias | Change from pre to 1 month post intervention
  "Blame" subscore of Anti-fat Attitudes Test, higher score means more bias

SECONDARY OUTCOMES:
Change in "Social" explicit bias | Change from pre to immediately post intervention (1 hour)
  "Social" subscore of Anti-fat Attitudes Test, higher score means more bias
Change in "Social" explicit bias | Change from pre to 1 month post intervention
  "Social" subscore of Anti-fat Attitudes Test, higher score means more bias
Change in "Physical" explicit bias | Change from pre to immediately post intervention (1 hour)
  "Physical" subscore of Anti-fat Attitudes Test, higher score means more bias
Change in "Physical" explicit bias | Change from pre to 1 month post intervention
  "Physical" subscore of Anti-fat Attitudes Test, higher score means more bias
Change in Implicit Bias | Change from pre to immediately post intervention (1 hour)
  Category of bias from Weight Implicit Association Test; Categories 1-4, higher category means more bias
Change in Implicit Bias | Change from pre to 1 month post intervention
  Category of bias from Weight Implicit Association Test; Categories 1-4, higher category means more bias

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We have a primary and secondary analysis planned for these data, once they are both published we will share the data within 6 months time via ICSPR database.
Supporting Information: Study Protocol
Time Frame: Within 6 months of publication, data will be available.
Access Criteria: Public Access Database.
URL: https://www.icpsr.umich.edu/icpsrweb/